CLINICAL TRIAL: NCT05630664
Title: Prospective Observational Study for the Implementation of Liquid Biopsy in the Follow-up of Patients With High-grade Gliomas and Meningiomas
Brief Title: Liquid Biopsy in High-grade Gliomas and Meningiomas
Acronym: SOPRANO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Alleanza Contro il Cancro (Other)
Responsible Party: Principal Investigator, Gaetano Finocchiaro, MD, IRCCS San Raffaele
Other Study IDs: ACCSOPRANO-22
Record Dates: First submitted 2022-09-14; First posted 2022-11-30 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: High Grade Glioma; High Grade Meningioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The general objective of this project is to evaluate the value of cell-free DNA circulating in plasma as a marker of tumor evolution in patients with high-grade gliomas and meningiomas.

To this end, we propose to longitudinally collect four samples of plasma at the following time points:

* T0: before surgery;
* T1: one month after surgery;
* T2: one month after the end of radiotherapy;
* T3 at the time of radiological progression.

The goal is to evaluate whether changes in plasma concentration of circulating cell-free DNA can help predict progression-free survival, overall survival, and response to therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Finding, on an MRI scan of the brain with gadolinium, of a brain lesion compatible with a primary brain tumor, intra- or extra-axial, suspected for a high-grade glioma or a high-grade meningioma, manifested with new onset neurological symptoms
* Clinical indication to perform a biopsy or surgical resection of the lesion
* Karnofsky Performance Status (KPS) ≥ 60
* Signature of informed consent

Exclusion Criteria:

* Absolute contraindications to magnetic resonance imaging or to the administration of gadolinium (e.g. patients with pacemakers or other non-magneto-compatible devices)
* Known positivity for HIV, HCV or HBV
* There are clinical, biological or instrumental data suggesting that the brain lesion is non-neoplastic in nature (e.g., abscess, vascular malformation, inflammatory disease of the Central Nervous System)
* Women who are pregnant or breastfeeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients with a newly diagnosed brain lesion compatible with high-grade glioma or high-grade meningioma, for whom a brain biopsy or exeresis has been indicated. Patients of both sexes, aged between 18 and 85 years-old, with a Karnofsky Performance Status (KPS)≥ 60 will be enrolled.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
cfDNA correlation with PFS | 1-3 days before surgery until disease progression (or at month 12 after surgery in the absence of disease progression)
  To evaluate whether circulating free DNA concentration in plasma at diagnosis correlates with progression-free survival.

SECONDARY OUTCOMES:
cfDNA correlation with OS | 1-3 days before surgery until patient death (or at month 12 if patient is alive)
  To valuate whether the concentration of circulating free DNA in plasma at the time of diagnosis correlates with overall survival
correlation between change in cfDNA concentration after surgery and PFS and OS | from day 30 (+/- 3 days) after surgery until disease progression, patient death (or at month 12 after surgery in the absence of disease progression)
  To evaluate whether a reduction in plasma concentration of circulating free DNA compared to preoperative values (T0) is seen one month after the surgical procedure (T1) and if this reduction is predictive of progression-free survival and overall survival.
correlation between change in cfDNA concentration one month after radiotherapy completion and tumor volume changes, as well as clinical status changes | values assessed at month 3.5 after surgery (+/- one week) compared with values assessed 1-3 days before surgery
  To evaluate, one month after the completion of radio (chemo) therapy (T2), the plasma concentration of circulating free DNA with respect to the pre-treatment values (T1), correlating with the volumetric and radiomic variations of the tumor in the magnetic resonance images (FLAIR sequence and T1 after injection of contrast medium), as well as with the changes in the patient's neurological status measured by the NANO score (Nayak et al., 2017) at the same timepoints.
cfDNA concentration changes at progression | values at the time of suspected radiological progression (or at month 12 in the absence of suspected radiological progression) compared with values assessed at month 3.5 after surgery (+/- one week)
  To evaluate at the time of suspected radiological progression (T3) the plasma concentration of circulating free DNA and its variations compared to the values detected one month after the end of radio (chemo) therapy (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Finocchiaro, MD, Principal Investigator — Ospedale San Raffaele, Milano, Italy
Locations (5):
- Italy (5):
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Istituto Clinico Humanitas IRCCS, Rozzano, MI
  - Istituto Oncologico Veneto, Padua, PD
  - Istituto Nazionale Tumori Regina Elena, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM